CLINICAL TRIAL: NCT00745290
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Group, Active Control Study to Evaluate the Safety and Efficacy of a Single Intraoperative Administration of SKY0402 For Prolonged Postoperative Analgesia in Subject Undergoing Total Knee Arthroplasty
Brief Title: A Phase 3 Study to Evaluate the Safety and Efficacy of SKY0402 in Subjects Undergoing Total Knee Arthroplasty
Acronym: TKA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SIMPLE TKA 311
Record Dates: First submitted 2008-08-29; First posted 2008-09-03 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-07

CONDITIONS: Postoperative Pain
Keywords: Total knee arthroplasty; Pain; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine HCl (Active Comparator): Single dose of 200 mg bupivacaine HCl administered intraoperatively via local infiltration
  Interventions: Drug: Bupivacaine HCl
- SKY0402 (Other): Single dose of 600 mg SKY0402 (study drug) administered intraoperatively via local infiltration
  Interventions: Drug: SKY0402

INTERVENTIONS:
Drug: Bupivacaine HCl — 200 mg bupivacaine HCl
  Other Names: Marcaine
  Arms: Bupivacaine HCl
Drug: SKY0402 — 600 mg SKY0402 (study drug).
  Other Names: DepoBupivacaine
  Arms: SKY0402

SUMMARY:
The primary objective is to demonstrate that SKY0402 is superior when compared to bupivacaine HCl in the management of postoperative pain for patients undergoing total knee arthroplasty.

DETAILED DESCRIPTION:
The primary objective is to demonstrate the superiority of SKY0402, compared with bupivacaine HC1, with respect to the extent and duration of the analgesic effect achieved by a single intraoperative administration of the study drug via local infiltration in subjects undergoing total knee arthroplasty (TKA).

The secondary objectives are to evaluate additional efficacy parameters and characterize the safety profile of SKY0402 in comparison with bupivacaine HCl.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years of age at the Screening Visit.
2. Female subjects only: Postmenopausal, surgically sterile, or willing to use acceptable means of contraception for at least 30 days after surgery including any of the following: hormonal contraceptives (e.g., oral, injectable, implantable starting at least 30 days before study drug administration), effective double-barrier methods (e.g., condoms with spermicide), intrauterine device, lifestyle with a personal choice of abstinence, nonheterosexual lifestyle, or a strictly monogamous relationship with a partner who has had a vasectomy.
3. Scheduled to undergo primary unilateral TKA under general or spinal anesthesia.
4. American Society of Anesthesiology (ASA) Physical Classification System class 1-4.
5. Able and willing to comply with all study visits and procedures.
6. Able to speak, read, and understand the language of the informed consent form, study questionnaires, and other instruments used for collecting subject-reported outcomes, in order to enable accurate and appropriate responses to pain scales and other required study assessments.
7. Willing and capable of providing written informed consent.

Exclusion Criteria:

1. Pregnancy, nursing, or planning to become pregnant during the study or within one month after dosing.
2. Use of any of the following medications within the times specified before surgery:

   * Long-acting opioid medication within 3 days.
   * Any opioid medication within 24 hours.
3. Concurrent painful physical condition or concurrent surgery that may require analgesic treatment in the postoperative period for pain that is not strictly related to the surgical site being administered study drug (e.g., significant pain from other joints, chronic neuropathic pain, concurrent contralateral TKA, concurrent foot surgery, etc.), which have the potential to confound the postoperative study assessments.
4. Body weight less than 60 kilograms (~132 pounds).
5. Contraindication to any of the pain-control agents planned for postoperative use (e.g., acetaminophen, morphine, oxycodone, ketorolac).
6. Contraindication to epinephrine, such as concurrent administration of ergot-type drugs, monoamine oxidase (MAO) inhibitors or antidepressants of triptoline or imipramine types, conditions where the production or exacerbation of tachycardia could prove fatal (e.g., poorly controlled thyrotoxicosis or severe heart disease), or any other pathological conditions that might be aggravated by the effects of epinephrine.
7. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
8. Suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
9. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, may interfere with study assessments or compliance.
10. Current or historical evidence of any clinically significant disease or condition that, in the opinion of the Investigator, may increase the risk of surgery or complicate the subject's postoperative course.
11. Significant medical conditions or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to study drugs and procedures, and expose the subject to an unreasonable risk as a result of participating in this clinical trial, such as: debilitating diseases, acute illnesses, hypotension, partial or complete conduction block, impaired cardiac function, untreated hypertension, advanced arteriosclerotic heart disease, cerebral vascular insufficiency, pre-existing abnormal neurological or neuromuscular disease (e.g., epilepsy, myasthenia gravis), advanced liver disease, severe renal impairment, advanced diabetes, comorbid conditions associated with an immunocompromised status, such as blood dyscrasias, HIV/AIDS, or recent chemotherapy.

    In addition, the subject will be ineligible to receive study drug if he or she meets the following criterion during surgery:
12. Any clinically significant event or condition uncovered during surgery (e.g., excessive bleeding), which occurs before study drug administration, that might render the subject medically unstable or complicate the subject's postoperative course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Davis, RN, Study Director — Pacira Pharmaceuticals, Inc
Locations (19):
- United States (19):
  - West Alabama Research, Inc., Birmingham, Alabama
  - Horizon Research Group, Inc., Alabama Orthopaedic Clinic, Mobile, Alabama
  - Drug Research and Analysis Corporation, Montgomery, Alabama
  - Sun Health Research Institute, Core Institute, Sun City West, Arizona
  - Scripps, La Jolla, California
  - Accurate Clinical Trials, Inc., Laguna Hills, California
  - Physicans Clinical Research Corp., Laguna Hills, California
  - Cedars of Sinai Medical Center, Los Angeles, California
  - Atlanta Knee and Sports Medicine, Decatur, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Insall Scott Kelly Institute, New York, New York
  - CTMG, Inc., Greenville, North Carolina
  - Duke University Medical Center, Raleigh-Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Allegheny Pain Management, Altoona, Pennsylvania
  - Ilumina Clinical Associates, Johnstown, Pennsylvania
  - Research Associates of Jackson, Jackson, Tennessee
  - Texas Orthopedic Specialists, PA, Grapevine, Texas
  - Memorial Hermann City Hospital, Houston, Texas

REFERENCES:
- [Derived] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine HCl: randomized in a 1:1 ratio to receive 200 mg bupivacaine HCl and stratified by site and by modality.
- SKY0402: randomized in a 1:1 ratio to receive 600 mg SKY0402 (study drug) and stratified by site and by modality.
Period: Overall Study
Arm/Group | Bupivacaine HCl | SKY0402
Started | 123 | 122
Completed | 123 | 122
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine HCl | SKY0402 | Total
Number analyzed (Participants) | 123 | 122 | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 52 | 119
  >=65 years | 56 | 70 | 126
Age Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.4) | 66.8 (10.6) | 65.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 83 | 156
  Male | 50 | 39 | 89
Region of Enrollment [Number; unit: participants]
  United States | 123 | 122 | 245

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) With Activity (NRS-A) Pain Intensity Scores
Description: The subject's pain intensity was assessed with activity (NRS-A), while actively flexing the involved knee from the maximum extension point to the maximum flexion point possible. The subject responded to the following question, "On a scale of 0 to 10, where 0 = no pain and 10 = worst possible pain, how much pain did you have while bending your knee?"
Time Frame: through 72 hours post surgery
Population: Note: 245 subjects were randomized and received study drug and were included in the analyses.
Measure: Mean (Standard Deviation); unit: Units on a scale*hours
Arm/Group | Bupivacaine HCl | SKY0402
Number analyzed (Participants) | 123 | 122
Units on a scale*hours | 335 (113) | 359 (124)

2. Secondary Outcome: Number of Participants With Adverse Events Through 96 Hours and Serious Adverse Events Through 30 Days
Time Frame: through 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Bupivacaine HCl | SKY0402
Serious Adverse Events (participants affected / at risk) | 18/123 | 12/122
Other Adverse Events (participants affected / at risk) | 107/123 | 108/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine HCl (N=123) | SKY0402 (N=122)
Cellulitis (Infections and infestations) | 0 (0) | 3
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 3 | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 (0)
Sedation (Nervous system disorders) | 0 | 1 (1)
Syncope (Nervous system disorders) | 1 | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postprocedural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bupivacaine HCl (N=123) | SKY0402 (N=122)
Nausea (Gastrointestinal disorders) | 71 | 76
Constipation (Gastrointestinal disorders) | 47 | 56
Vomiting (Gastrointestinal disorders) | 42 | 38
Haemorrhagic anemia (Blood and lymphatic system disorders) | 8 | 4
Anemia postoperative (Injury, poisoning and procedural complications) | 10 | 12
Procedural pain (Injury, poisoning and procedural complications) | 9 | 10
Pyrexia (General disorders) | 16 | 14
Oedema peripheral (General disorders) | 5 | 9
Pruritis (Skin and subcutaneous tissue disorders) | 16 | 11
Insomnia (Psychiatric disorders) | 9 | 9
Dizziness (Nervous system disorders) | 3 | 8
Hypotension (Vascular disorders) | 4 | 9
Tachycardia (Cardiac disorders) | 3 | 7
Anemia (Blood and lymphatic system disorders) | 28 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No